CLINICAL TRIAL: NCT07346573
Title: A Retrospective Single-Center Study Utilizing AI-Based Radiomics on Pre- and Post-Radiotherapy CT Images to Explore the Safety Dose Threshold in Liver Malignancy Radiation Therapy
Brief Title: Radiotherapy Safety for Liver Malignancies Using Post-Treatment Imaging
Status: Completed | Type: Observational
Sponsor: Cao peiguo (Other)
Responsible Party: Sponsor-Investigator, Cao peiguo, Professor peiguo Cao, Chief Physician of Radiation Oncology Department, the Third Xiangya Hospital, The Third Xiangya Hospital of Central South University
Organization: The Third Xiangya Hospital of Central South University (Other)
Other Study IDs: CSU-2024-HCCRT001
Record Dates: First submitted 2025-12-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-05

CONDITIONS: Liver Neoplasms; Radiation-Induced Liver Injury
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FLR Group: Patients who developed Focal Liver Reaction (FLR) on follow-up CT imaging after radiotherapy
  Interventions: Other: Clinically Delivered Radiation Therapy (e.g., SBRT/IMRT) for Liver Cancer
- Non-FLR Group: Patients who did not develop Focal Liver Reaction (FLR) on follow-up CT imaging after radiotherapy
  Interventions: Other: Clinically Delivered Radiation Therapy (e.g., SBRT/IMRT) for Liver Cancer

INTERVENTIONS:
Other: Clinically Delivered Radiation Therapy (e.g., SBRT/IMRT) for Liver Cancer — This is a retrospective observational study. The intervention (radiotherapy) was administered as part of standard clinical care prior to the study. Researchers are analyzing the outcomes of this previously delivered intervention.

SUMMARY:
The goal of this retrospective observational study is to investigate the safety of radiation therapy for liver malignancies by analyzing data from patients who have already completed this treatment . The main questions it aims to answer are:

What is the specific radiation dose level that leads to a visible change on CT scans called a Focal Liver Reaction (FLR)? Why do some patients develop these imaging changes while others do not, based on their scan features and clinical information? Researchers will compare patients who developed FLR with those who did not to identify the factors associated with this reaction.

This study uses existing medical records and images; therefore, participants will not need to undergo any new interventions or procedures.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary liver malignancies, including hepatocellular carcinoma (HCC), intrahepatic cholangiocarcinoma (ICC), and secondary liver tumors.
* Liver function of Child-Pugh classification A or B.
* Completed EBRT treatment as planned.
* No other local treatment of liver lesions between EBRT and the follow-up imaging examination.
* Complete imaging re-examination data.
* Three-phase enhancement CT scans showing typical Focal Liver Reaction (FLR).
* The registration effect of follow-up CT and planning CT is satisfactory.

Exclusion Criteria:

* History of upper abdominal radiotherapy or liver transplantation.
* Failure to complete radiotherapy as scheduled.
* Previous cancer treatment-related toxicities that did not return to baseline or grade 0-1 (except for hair loss and peripheral neuropathy).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with primary or metastatic liver malignancies who received liver radiotherapy (e.g., SBRT or IMRT) at the Third Xiangya Hospital of Central South University between July 2015 and September 2024 , and had complete dosimetric data and follow-up CT imaging available for retrospective analysis.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Dose Threshold for Focal Liver Reaction (FLR) | Retrospectively, data collected from the beginning of radiotherapy to one year after the end of radiotherapy
  The minimum radiation dose (in Gy) required to induce a radiologically visible Focal Liver Reaction (FLR) on follow-up CT imaging, as assessed by CT scan.
Predictors of FLR Susceptibility | Retrospectively, data collected from the beginning of radiotherapy to one year after the end of radiotherapy
  Differences in radiomic features and clinical baseline characteristics (e.g., age, gender, liver function, and tumor size) between patients with radiologically confirmed Focal Liver Reaction (FLR) and those without, assessed by radiomic analysis and clinical data review.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No